CLINICAL TRIAL: NCT01231711
Title: Improving Quality-of-life and Depressive Symptoms for OEF/OIF Combat Veterans: Assessing the Benefits of Interactive, Internet-based Psychotherapy and Peer-to-peer Support
Brief Title: Improving Quality-of-life and Depressive Symptoms of Combat Veterans Via Internet-based Intervention
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prevail Health Solutions, LLC (Industry)
Collaborators: Rise Consulting, LLC (Unknown); McCormick Foundation (Unknown)
Responsible Party: Brock Hokenson, Operations Officer, Prevail Health Solutions, LLC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 24633-1
Record Dates: First submitted 2010-10-28; First posted 2010-11-01 (Estimated); Last update posted 2010-11-01 (Estimated); Status verified 2010-10

CONDITIONS: Depression; Post-Traumatic Stress Disorder; Functional Status
Keywords: depression; post traumatic stress syndrome; functional status; veteran; military; stigma; mental health self-efficacy
MeSH Terms: conditions — Depression; Stress Disorders, Post-Traumatic; Combat Disorders; Social Stigma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vets Prevail (Experimental): N=50. Participants were recent veterans (deployed after September 11, 2001) of operations in Iraq and Afghanistan who were experiencing depression/distress symptoms at the time of screening (CES-D > 8) but who were not considered to be inappropriate for a health promotion intervention (CES-D > 35 indicating severe depressed mood or exhibiting self-harm risk).
  Interventions: Behavioral: Vets Prevail

INTERVENTIONS:
Behavioral: Vets Prevail — The intervention has two primary components that are both delivered over the Internet:
  The first component is a structured series of brief peer-to-peer instant messaging "Chats" structured around ensuring effective motivation, engagement, and completion. This component was modeled after Motivational Interviewing (MI) techniques. The peer-to-peer contact was provided by a master's level social worker, as well as by trained and certified combat veterans who completed the Vet-to-Vet counseling certificate program offered by the Depression and Bipolar Support Alliance (DBSA).
  The second component consists of six 30-minute "e-Learning Lessons" using standard Cognitive Behavioral Therapy (CBT) approaches to reducing depressive and anxiety symptoms and strengthening coping skills.
  Other Names: Warriors Prevail

SUMMARY:
Background: Current military involvement in Afghanistan (Operation Enduring Freedom - OEF) and Iraq (Operation Iraqi Freedom - OIF) has created unforeseen burdens on the mental health and well-being of US service women and men. Although OEF/OIF service members and veterans are at high risk of developing sub-threshold combat stress and depressive symptoms or full disorders in the post-deployment period, only a small fraction ever receive care. The VETS PREVAIL Intervention, which combines Cognitive-Behavioral-Therapy-based (CBT-based) coping skills training with peer-to-peer support and counseling, was specifically designed to offer the returning OEF/OIF service member or veteran an accessible and confidential first step to care.

Evaluation Study: RISE Consulting, lead by Dr. Benjamin W. Van Voorhees, MD, MPH, was contracted to supervise a pilot study of potential benefit, feasibility and safety of the VETS PREVAIL Intervention. The study would consist of a single group pre/post comparison study of N=50 recent OEF/OIF veterans in the frame work of a phase 1 clinical trial (phase 1). Feasibility (adherence and satisfaction), evidence of clinical benefit would be evaluated through changes in the following clinical self-report measures: i) symptoms of depressed mood (Center for Epidemiologic Studies Depression Scale, CES-D), ii) post traumatic stress disorder (Post Traumatic Stress Disorder Checklist-Military, PCL-M), and iii) functional status (Short Form 12, SF-12), as well as changes in key attitudes toward mental health care seeking (intent to seek treatment, mental health self-efficacy and stigma).

DETAILED DESCRIPTION:
Intervention overview content and design:

The intervention, VETS PREVAIL, will empower the user to gain control over life problems through enhancement of coping strategies, self-care, social support, and a repertoire of problems solving skills in an interactive internet intervention. This intervention will have two components: internet delivery of the intervention and brief person-to-person electronic contact structured around ensuring effective motivation, engagement, and completion. The coaching model for the person-to-person contact will be based on motivational interviewing with masters level social workers , as well as contact with peers who have completed the Vet-to-Vet certificate program offered by the Depression and Bipolar Support Alliance (DBSA). The internet component is focused on combat stress, self-assessment, coping strategies, problem solving, and social support.

Trainer Role:

During the 6 weeks of Vets Prevail a trainer, a masters level social worker, will engage with subjects through one online chat per week, post lesson (approximately 15 minute time blocks; duration will vary per subject). The total amount of person-to-person contact time, with a trainer, is an estimated 90 minutes throughout the 6 week program; contact time may vary per subject. The trainer will use motivational interviewing to clarify concepts within each week's lesson. In addition, the trainer will be responsible for making referrals and follow ups, when needed.

Masters level social work education trains people to use evidence-based knowledge derived from research, practice evaluation and theories of human development and behavior and social systems to analyze complex situations between individuals and their environment, in addition to facilitating individual, organizational, social and cultural changes.

Peer Role:

During the 6 weeks of Vets Prevail a peer, a DBSA certified veteran, will engage with subject through one online chat per week, pre lesson (approximately 15 minute time blocks: duration will vary per subject). The total amount of person-to-person contact time, with a peer, is an estimated 60 minutes throughout the 6 week program; contact time my vary per subject. The purpose of the peer engagement is to motivate the subject to complete the activities they schedule for themselves during the week and to apply the lessons from each session into their lives.

DBSA training trains people to use their experiences to work with others. Training features a nationally-developed recovery philosophy curriculum to enhance wellness and treatment strategies, through peer delivery services.

Internet based component:

The current intervention will have four major sections. The first section will relate stress in the context of depressive symptoms with direct tactics that can be immediately implemented to reduce symptoms and guide users towards their individual goals. The second section will demonstrate how to recognize treatment obstacles and organizing implementation of the tactics from section one. The third section addresses overcoming treatment obstacles along with reinforcing reduction of symptoms and goal-directed action. The fourth section provides instruction and application of personal problem-solving, taking goal-directed action to full implementation. The intervention concludes with a review, a reinforcement of personally-relevant treatment applications, and an evaluation of techniques. The internet component will also require active engagement of the individual with interactive activities to improve learning/skill building along with other activities designed to identify how they would manage specific behavioral symptoms (skill development). The internet component will consist of 6 individual sessions, with approximately one week between sessions. The electronic chat with the peer will occur directly before the subjects view this content, and the chat with the trainer occurs immediately afterwards so the trainer can answer any questions about the content the subject might have.

ELIGIBILITY:
Inclusion Criteria:

* >=18 years of age
* A veteran of the U.S. military having served in the Iraq or Afghanistan theaters in the last 5 years.
* CES-D(20) score >8
* Access to high-speed internet
* Own a cell phone with text message capability
* speak and read the English language

Exclusion Criteria:

* psychiatric hospitalizations within past 10 years
* any past suicide attempt
* diagnoses of schizophrenia or bipolar disorder
* CES-D(20) score >36
* discontinued or altered dosage of medication within 10 days prior to enrollment
* score >=2 on the alcohol/drug assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-09; Primary Completion 2010-02 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Center for Epidemiologic Studies Depression Scale 10 (CES-D 10) | baseline, 4 weeks, 8 weeks, 12 weeks
  The Center for Epidemiologic Studies Depression Scale (CES-D) is one of the most common screening tests for helping an individual to determine his or her depression quotient. The quick self-test measures depressive feelings and behaviours during the past week.

SECONDARY OUTCOMES:
Post Traumatic Stress Disorder Checklist-Military (PCL-M) | baseline, week 4, week 8, week 12
  The PTSD Checklist-Military (PCL-M) is a 17-item self-report measure of PTSD symptoms that requires respondents to rate the severity of each symptom during the past 30 days on a five-point ordinal scale. A total PCL-M score was created by summing the item ratings.
12-Item Short Form Health Survey (SF-12) | baseline, week 4, week 8, week 12
  The SF-12 is a generic measure and does not target a specific age or disease group. It is a shorter, valid alternative to the SF-36. The SF-12 is weighted and summed to provide separate scales for an individuals phisical and mental health called the Physical Composite Score (PCS) and Mental Composite Score (MCS).

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin VanVoorhees, MD, MPH, Principal Investigator — Rise Consulting, LLC; Brock K Hokenson, MBA, Study Director — Prevail Health Solutions
Locations (1):
- Prevail Health Solutions, Chicago, Illinois, United States